CLINICAL TRIAL: NCT05134558
Title: Xenon-enhanced Ventilation CT-guided Radiotherapy for Lung Cancer Treatment: Functional Protection of the Lung and Prevention of Radiation Pneumonitis
Brief Title: Xenon-enhanced Ventilation CT-guided Radiotherapy for Lung Cancer Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201912128RIN
Record Dates: First submitted 2021-09-22; First posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-09

CONDITIONS: Lung Cancer; Radiation Therapy Complication
Keywords: lung cancer; Radiation Therapy; Xenon-enhanced ventilation CT
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Xenon-enhanced Ventilation CT-guided Radiotherapy (Experimental): Patients will be receiving Xenon-enhanced Ventilation CT-guided Radiotherapy for functional lung avoidance. The doses for the tumors, lungs, and organs at risk will be examined and evaluated.
  Interventions: Radiation: Xenon-enhanced Ventilation CT-guided Radiotherapy

INTERVENTIONS:
Radiation: Xenon-enhanced Ventilation CT-guided Radiotherapy — Xenon-enhanced Ventilation CT-guided Radiotherapy for functional protection of the lung

SUMMARY:
The investigators aim to use xenon-enhanced ventilation computed tomography (CT) to design personalized functional lung avoidance radiotherapy for lung cancer patients who are scheduled to receive lung radiation therapy. The investigators' goal is to optimally protect the lung function of the patients and reduce the incidence of radiation pneumonitis.

DETAILED DESCRIPTION:
There has been an increase in the application of radiation therapy in the treatment of lung tumors; however, the associated side effect, called radiation pneumonitis, can significantly reduce lung function and the quality of life of patients, eventually leading to fatal consequences. The investigators aim to use xenon-enhanced ventilation computed tomography (CT) to design personalized functional lung avoidance radiotherapy for lung cancer patients who are scheduled to receive lung radiation therapy. The investigators' goal is to optimally protect the lung function of the patients and reduce the incidence of radiation pneumonitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20-80 years, with lung cancer receiving thoracic radiotherapy in NTUH, from February 2020 to December 2024.

Exclusion Criteria:

* The age is less than 20 years old or older than 80 years old.
* Unstable clinical condition, unable to maintain apnea for 15 second, and history of prior adverse reaction to xenon.
* Renal insufficiency patients.
* Claustrophobia
* Those who are pregnant.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-02-04 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of radiation pneumonia | Within 1 year of radiation therapy
  Incidence of radiation pneumonia

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided